CLINICAL TRIAL: NCT03294590
Title: Randomized Controlled Trial of Interactive Parent-Targeted Text Messaging in Pediatric Clinics to Reduce Caries Among Urban Children
Brief Title: Interactive Parent-Targeted Text Messaging in Pediatric Clinics to Reduce Caries Among Urban Children
Acronym: iSmile
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H-36857; 4UH3DE025492-03 (NIH)
Record Dates: First submitted 2017-09-21; First posted 2017-09-27 (Actual); Results first posted 2023-05-18 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Caries, Dental; Health Behavior
Keywords: Child oral health behaviors; Text messages; Motivation; Self efficacy; Outcome Expectations; Sugar sweetened beverage consumption; Fluoride varnish; Healthy eating; Parent oral health behaviors; Parent oral health attitudes; Fluoride; early childhood caries
MeSH Terms: conditions — Dental Caries; Health Behavior

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Outcome Assessors and Oral Health Examiners will be blind to treatment condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral health text messages (OHT) (Experimental): Participants in this arm will receive the OHT parent targeted text messages to reduce caries and improve oral health behaviors among low income families visiting community-based, urban pediatric clinics.
  Interventions: Other: OHT Parent targeted text messages
- Child wellness text messages (CWT) (Active Comparator): Participants in this arm will receive the CWT parent targeted text messages to improve child wellness (e.g., reading time, safety) among low income families visiting community-based, urban pediatric clinics.
  Interventions: Other: CWT Parent targeted text messages

INTERVENTIONS:
Other: OHT Parent targeted text messages — For the Oral health text message (OHT) group, the parent targeted text messaging program will include two core topics and a menu of options to choose from, all of which pertain to oral health.
  Arms: Oral health text messages (OHT)
Other: CWT Parent targeted text messages — For the CWT group, the parent targeted text messaging program will include two core topics and a menu of options to choose from, all of which pertain to child wellness.
  Arms: Child wellness text messages (CWT)

SUMMARY:
This is a randomized clinical trial to test the efficacy of a parent-targeted text message-based intervention program on caries incidence and oral health behaviors (child and parent). Parents (n= 850) across all pediatric clinic sites (Boston Medical Center and Community Health Centers (CHCs); DotHouse CHC, South End Community Health Center, and Codman Square CHC) will be randomized to receive either text messages (TMs) regarding oral health or TMs regarding child wellness. The study will enroll English and Spanish speaking parents and their youngest child who is < 7 years old, has at least one tooth showing, and attends the targeted pediatric clinic to receive primary care (n= 1700). Parents will complete self-report surveys at baseline, and 2, 4, 12, and 24-months after baseline; receive and respond to TM assessments during the 4-month intervention; and will also receive TMs during a 'booster' period of one month, which will occur 12-months post baseline. Parent's children will be assessed for caries by a clinical oral examination performed by licensed Clinical Examiners at baseline, 12-and-24-months post-baseline.

ELIGIBILITY:
Inclusion Criteria: Caregiver and child must meet all of the following:

1. Caregiver must be a parent or legal guardian of a child less than 7 years old, and the child must have their first tooth showing
2. The child must receive medical care at one of the participating pediatric clinics.
3. Speak, understand, and read either English or Spanish
4. Have a mobile phone.

Exclusion Criteria: If the caregiver or child meets any of the following criteria, the dyad will be excluded from participation in this study

1. Children with severe congenital tooth malformations: At screening the caregiver will be asked if their child has known systemic diseases associated with abnormal tooth development or abnormal oral health status such as cleft lip or palate, amelogenesis imperfecta, or dentinogenesis imperfecta.
2. Children who cannot complete the baseline oral health exam.

Ages: 0 Months to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 754 (Actual)
Dates: Start 2018-03-09 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Belinda Borrelli, PhD, Principal Investigator — Henry M. Goldman School of Dental Medicine
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Borrelli B, Endrighi R, Heeren T, Adams WG, Gansky SA, Werntz S, Rueras N, Stephens D, Ameli N, Henshaw MM. Parent-Targeted Oral Health Text Messaging for Underserved Children Attending Pediatric Clinics: A Randomized Clinical Trial. JAMA Netw Open. 2025 Jan 2;8(1):e2452780. doi: 10.1001/jamanetworkopen.2024.52780. PMID 39745701

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 754 dyads (parents or caregivers and child) were enrolled and randomized.
Period: Overall Study
Arm/Group | Oral Health Text Messages (OHT) | Child Wellness Text Messages (CWT)
Started (Number of parent/caregiver-child dyads randomized) | 377 | 377
Number of Parent/Caregiver Participants | 377 | 377
Number of Children Participants | 377 | 377
4-month Time Point (Survey) | 290 (Number of parents/caregivers completing the 4-month questionnaire assessment) | 288 (Number of parents/caregivers completing the 4-month questionnaire assessment)
12-month Time Point (Survey) | 282 (Number of parents/caregivers completing the 12-month questionnaire assessment) | 290 (Number of parents/caregivers completing the 12-month questionnaire assessment)
12-month Time Point (Oral Exam) | 206 (Number of children completing the 12-month oral health exam) | 185 (Number of children completing the 12-month oral health exam)
24-month Time Point (Survey) | 272 (Number of parents/caregivers completing the 24-month questionnaire assessment) | 270 (Number of parents/caregivers completing the 24-month questionnaire assessment)
24-month Time Point (Oral Exam) | 160 (Number of children completing the 24-month oral health exam) | 156 (Number of children completing the 24-month oral health exam)
Completed (542 parent/caregiver participants completed at least the questionnaire assessment of the final study visit (24-month time point)) | 272 | 270
Not Completed | 105 | 107
Not completed — Lost to Follow-up | 105 | 107

BASELINE CHARACTERISTICS:
Population: 754 parent/caregiver-child dyads were assessed for baseline measures (total 1,508 participants)
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Health Text Messages (OHT) | Child Wellness Text Messages (CWT) | Total
Number analyzed (Participants) | 754 | 754 | 1508
Age, Continuous [Mean (Standard Deviation); unit: years] — Mean age of parent/caregiver and children participants Population: 754 Parent/caregiver-child dyads were assessed for baseline measures for a total of 1,508 participants
  years
    Parent/caregiver participants: number analyzed (Participants) | 377 | 377 | 754
    Parent/caregiver participants | 32.8 (7.0) | 33.0 (7.4) | 32.9 (7.2)
    Children participants: number analyzed (Participants) | 377 | 377 | 754
    Children participants | 2.9 (1.7) | 2.8 (1.6) | 2.9 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Sex of parent/caregiver and children participants Population: 754 Parent/caregiver-child dyads were assessed for baseline measures for a total of 1,508 participants
  Participants
    Parent/caregiver participants: number analyzed (Participants) | 377 | 377 | 754
    Parent/caregiver participants: Female | 358 | 355 | 713
    Parent/caregiver participants: Male | 19 | 22 | 41
    Children participants: number analyzed (Participants) | 377 | 377 | 754
    Children participants: Female | 186 | 191 | 377
    Children participants: Male | 191 | 186 | 377
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity of parent/caregiver and children participants Population: 754 Parent/caregiver-child dyads were assessed for baseline measures for a total of 1,508 participants
  Participants
    Parent/caregiver participants: number analyzed (Participants) | 377 | 377 | 754
    Parent/caregiver participants: Hispanic or Latino | 98 | 96 | 194
    Parent/caregiver participants: Not Hispanic or Latino | 270 | 270 | 540
    Parent/caregiver participants: Unknown or Not Reported | 9 | 11 | 20
    Children participants: number analyzed (Participants) | 377 | 377 | 754
    Children participants: Hispanic or Latino | 114 | 113 | 227
    Children participants: Not Hispanic or Latino | 252 | 251 | 503
    Children participants: Unknown or Not Reported | 11 | 13 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race of parent/caregiver and children participants Population: 754 Parent/caregiver-child dyads were assessed for baseline measures for a total of 1,508 participants
  Participants
    Parent/caregiver participants: number analyzed (Participants) | 377 | 377 | 754
    Parent/caregiver participants: American Indian or Alaska Native | 2 | 1 | 3
    Parent/caregiver participants: Asian | 7 | 9 | 16
    Parent/caregiver participants: Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
    Parent/caregiver participants: Black or African American | 235 | 205 | 440
    Parent/caregiver participants: White | 46 | 48 | 94
    Parent/caregiver participants: More than one race | 25 | 39 | 64
    Parent/caregiver participants: Unknown or Not Reported | 61 | 73 | 134
    Children participants: number analyzed (Participants) | 377 | 377 | 754
    Children participants: American Indian or Alaska Native | 2 | 1 | 3
    Children participants: Asian | 6 | 4 | 10
    Children participants: Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
    Children participants: Black or African American | 225 | 199 | 424
    Children participants: White | 33 | 41 | 74
    Children participants: More than one race | 58 | 72 | 130
    Children participants: Unknown or Not Reported | 52 | 59 | 111
Region of Enrollment [Number; unit: participants]
  United States | 754 | 754 | 1508

OUTCOME MEASURES:

1. Primary Outcome: Dental Caries Increment
Description: Surface level caries data in children was collected by calibrated clinical examiners (blind to treatment condition), utilizing the OHDC Modified ICDAS methodology, will allow calculation of caries increment (development of a new cavitated lesion or filled surface on a previously sound tooth surface).
Time Frame: 24-month time point (oral assessment)
Population: Number of children with any new dental caries in primary teeth (using multiple imputation methods to account for missing oral health assessment data at 24-month)
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Health Text Messages (OHT) | Child Wellness Text Messages (CWT)
Number analyzed (Participants) | 377 | 377
Participants | 162 | 161

2. Primary Outcome: Parent/Caregiver Confidence to Brush
Description: 9-item self-efficacy measure to assess parent/caregiver participant confidence in their ability to brush their child's teeth under different situations. (Finlayson measure; range 1 - 4; higher scores mean better outcome)
Time Frame: 4-month time point (survey)
Population: Scores on a self-efficacy measure (range 1 - 4; higher scores mean better outcome)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oral Health Text Messages (OHT) | Child Wellness Text Messages (CWT)
Number analyzed (Participants) | 290 | 288
score on a scale | 2.9 (1.2) | 2.8 (1.2)

3. Primary Outcome: Parent/Caregiver Motivation to Perform Oral Health Behaviors
Description: A oral health motivation measure to assess parent/caregiver participants motivation to engage in recommended child oral health behaviors (score range 1 - 7; higher scores mean better outcome)
Time Frame: 4-month time point (survey)
Population: Scores on a motivation measure (range 1 - 7; higher scores mean better outcome)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oral Health Text Messages (OHT) | Child Wellness Text Messages (CWT)
Number analyzed (Participants) | 290 | 288
score on a scale | 6.2 (1.2) | 6.0 (1.3)

4. Primary Outcome: Parent/Caregiver Outcome Expectations for Oral Health Behaviors
Description: An outcome expectancies measure to assess the degree to which parent/caregiver participants perceive that performing the oral health behaviors (e.g., brushing) will lead to the desired outcome (e.g., reduced dental caries) in their children (Stewart et al., 1997; range 1 - 4; higher scores mean better outcome).
Time Frame: 4-month time point (survey)
Population: Scores on an outcome expectancies measure (range 1 - 4; higher scores mean better outcome)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oral Health Text Messages (OHT) | Child Wellness Text Messages (CWT)
Number analyzed (Participants) | 290 | 288
score on a scale | 3.69 (0.67) | 3.68 (0.60)

5. Primary Outcome: Self-efficacy to Perform Oral Health Behaviors
Description: The overall self-efficacy score represents how sure parent/caregiver participants are that they can engage in recommended behavior to take care of their children's teeth. (Based on Albino et al 2017; range 1 - 7; higher scores mean better outcome).
Time Frame: 4-month time point (survey)
Population: Scores on a confidence (self-efficacy) measure (range 1 - 7; higher scores mean better outcome)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oral Health Text Messages (OHT) | Child Wellness Text Messages (CWT)
Number analyzed (Participants) | 290 | 288
score on a scale | 6.3 (1.1) | 6.2 (1.2)

6. Primary Outcome: Dental Caries Increment (Surface Level)
Description: Caries data in children participants collected by calibrated clinical examiners (blind to treatment condition), utilizing the OHDC Modified ICDAS methodology, will allow calculation of a surface of tooth-level caries increment (development of a new cavitated lesion or filled surface on a previously sound tooth surface).
Time Frame: 24-month time point (oral assessment)
Population: Number of tooth surfaces with new caries in children participants
Measure: Count of Units; unit: Tooth surfaces
Units Other Than Participants: Tooth surfaces
Arm/Group | Oral Health Text Messages (OHT) | Child Wellness Text Messages (CWT)
Number analyzed (Participants) | 160 | 156
Number analyzed (Tooth surfaces) | 13553 | 13477
Tooth surfaces | 545 | 496

7. Secondary Outcome: Text Message Program Length Satisfaction
Description: One item adapted from the Mobile App Rating Scale (MARS) to measure parent/caregiver participants satisfaction with the duration of the text message program.
Time Frame: 4-month time point (survey)
Population: The iSmile study consisted of "oral health" text messages for parent/caregiver participants in the OHT arm, and "child wellness" text messages for parent/caregiver participants in the CWT arm. Text message program length satisfaction assessed the number of parent/caregiver participants who selected each response option to: "You've been receiving the iSmile text messages for about four months. What do you think about the length of the program?"
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Health Text Messages (OHT) | Child Wellness Text Messages (CWT)
Number analyzed (Participants) | 290 | 288
Participants
  It was just about right | 193 | 172
  The program should last longer | 68 | 80
  The program should be shorter | 29 | 36

8. Secondary Outcome: Parents' Perceived Impact of iSmile
Description: Three items adapted from the MARS to measure the perceived impact of the OHT text message program on parent/caregiver participants' attitudes towards their child's oral health (range 1 - 7; higher scores mean a better outcome).
Time Frame: 4-month time point (survey)
Population: Parent/caregiver participants in the OHT arm responded to "How much do you think iSmile had a positive impact on?".. (1='not at all' to 7='very much'; higher scores mean a better outcome)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- OHT Group: Subjects receive oral health text messages (brushing, visiting the dentist, fluoride, reducing sugar sweetened beverages and healthy eating, bedtime routing, and bottle/sippy cup use)
Arm/Group | OHT Group
Number analyzed (Participants) | 290
units on a scale
  Making sure your child's teeth are brushed | 6.4 (1.3)
  Decreasing the amount of sugar-sweetened beverages your child drinks | 5.9 (1.8)
  Your feelings on taking your child to the dentist | 6.1 (1.6)

9. Secondary Outcome: Child Preventive Dental Visits
Description: One item adapted from the Basic Research Factors Questionnaire (BRFQ) to assess the number of parent/caregiver participants who indicated that their child had a preventive dental visit.
Time Frame: 4-month, 12-month, and 24-month time points (survey)
Population: Number of parent/caregiver participants who indicated that their child had a preventive dental visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Health Text Messages (OHT) | Child Wellness Text Messages (CWT)
Number analyzed (Participants) | 377 | 377
Participants
  24-month: number analyzed (Participants) | 272 | 270
  24-month | 207 | 181
  12-month: number analyzed (Participants) | 282 | 290
  12-month | 180 | 157
  4-month: number analyzed (Participants) | 290 | 288
  4-month | 162 | 131

10. Secondary Outcome: Fluoridated Toothpaste Use
Description: One item derived from the Basic Research Factors Questionnaire (BRFQ) to measure whether parent/caregiver participants use toothpaste containing fluoride when brushing their child's teeth.
Time Frame: 4-month, 12-month, and 24-month time points (survey)
Population: Number of parent/caregiver participants indicating use of fluoridated toothpaste to brush their child's teeth.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Health Text Messages (OHT) | Child Wellness Text Messages (CWT)
Number analyzed (Participants) | 377 | 377
Participants
  24-month: number analyzed (Participants) | 272 | 270
  24-month | 225 | 207
  12-month: number analyzed (Participants) | 282 | 290
  12-month | 229 | 215
  4-month: number analyzed (Participants) | 290 | 288
  4-month | 225 | 210

11. Secondary Outcome: Perceived Impact of OHT Program on Parental Awareness
Description: One item adapted from the Basic Research Factors Questionnaire (BRFQ) to measure parent/caregiver participants' (in the OHT arm) awareness of their child oral health.
Time Frame: 24-month (survey)
Population: Number of parent/caregiver participants in the OHT arm endorsing each response category in response to: "iSmile has increased my awareness of my child's oral health (1='strongly disagree, to 5='strongly agree')
Measure: Count of Participants; unit: Participants
Groups:
- OHT Group: Subjects received oral health text messages (brushing, visiting the dentist, fluoride, reducing sugar sweetened beverages and healthy eating, bedtime routing, and bottle/sippy cup use)
Arm/Group | OHT Group
Number analyzed (Participants) | 272
Participants
  1 - strongly disagree | 7
  2 - | 3
  3 - | 14
  4 - | 33
  5 - strongly agree | 207
  prefer not to answer | 8

12. Secondary Outcome: Child Diet - Food Frequency
Description: Parent/caregiver participants completed a food frequency questionnaire (FFQ) to assess their child's diet. Food/beverages items in the FFQ are categorized into groups according to the degree to which they promote dental caries, and a weighted estimated cariogenicity score (ECS) is computed (minimum and maximum scores range 0 - 3.80; higher scores mean a worse outcome).
Time Frame: 4-month, 12-month, and 24-month time points (survey)
Population: The estimated cariogenic score derived from a food frequency questionnaire (higher scores mean a worse outcome).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oral Health Text Messages (OHT) | Child Wellness Text Messages (CWT)
Number analyzed (Participants) | 377 | 377
score on a scale
  24-month: number analyzed (Participants) | 272 | 270
  24-month | 2.22 (0.31) | 2.27 (0.27)
  12-month: number analyzed (Participants) | 282 | 290
  12-month | 2.23 (0.30) | 2.23 (0.24)
  4-month: number analyzed (Participants) | 290 | 288
  4-month | 2.18 (0.28) | 2.22 (0.24)

13. Secondary Outcome: Child Diet - Beverage Intake
Description: Parent/caregiver participants completed the beverage questionnaire for preschoolers (BEVQ-PS) to assess their child's beverage intake. For each beverage item, the frequency and the amount of consumption are computed as average fluid ounces per day, and a composite score is computed for sugar sweetened beverages (including 100% fruit juice) consumption and then categorized into higher consumption (vs lower).
Time Frame: 4-month, 12-month, and 24-month time points (survey)
Population: Number of parent/caregiver participants indicating that their child consumed higher sugar sweetened beverages including 100% fruit juice (="more than 4.5 fluid ounces per day").
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Health Text Messages (OHT) | Child Wellness Text Messages (CWT)
Number analyzed (Participants) | 377 | 377
Participants
  24-month: number analyzed (Participants) | 272 | 270
  24-month | 125 | 142
  12-month: number analyzed (Participants) | 282 | 290
  12-month | 145 | 131
  4-month: number analyzed (Participants) | 290 | 288
  4-month | 128 | 141

14. Secondary Outcome: Child Tooth Brushing
Description: An investigator-developed composite measure derived from the number of days and number of times parent/caregiver participants brushed or supervised brushing their child's teeth during a week (range: 0 - 21; higher scores mean a better outcome).
Time Frame: 4-month, 12-month, and 24-month time points (survey)
Population: Number of child tooth brushings per week (range: 0 - 21; higher scores mean a better outcome)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oral Health Text Messages (OHT) | Child Wellness Text Messages (CWT)
Number analyzed (Participants) | 377 | 377
units on a scale
  24-month: number analyzed (Participants) | 272 | 270
  24-month | 12.0 (4.5) | 11.1 (5.1)
  12-month: number analyzed (Participants) | 282 | 290
  12-month | 12.0 (4.4) | 11.6 (4.6)
  4-month: number analyzed (Participants) | 290 | 288
  4-month | 12.9 (3.7) | 11.3 (5.0)

15. Secondary Outcome: Parent/Caregiver Tooth Brushing
Description: An investigator-developed composite measure derived from the number of days and number of times parent/caregiver participants brushed their teeth during a week (range: 0 - 21; higher scores mean a better outcome).
Time Frame: 4-month, 12-month, and 24-month time points (survey)
Population: Number of parent/caregiver participants tooth brushings per week (range: 0 - 21; higher scores mean a better outcome).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oral Health Text Messages (OHT) | Child Wellness Text Messages (CWT)
Number analyzed (Participants) | 377 | 377
units on a scale
  24-month: number analyzed (Participants) | 272 | 270
  24-month | 12.7 (3.8) | 12.3 (4.5)
  12-month: number analyzed (Participants) | 282 | 290
  12-month | 12.7 (4.2) | 12.5 (4.4)
  4-month: number analyzed (Participants) | 290 | 288
  4-month | 13.1 (3.8) | 12.4 (4.2)

16. Secondary Outcome: Child Oral Health-related Quality of Life
Description: The Early Childhood Oral Health Impact Scale (ECOHIS) to measure parent/caregiver participants' perceptions of their child's oral health (range 0 - 16; higher scores mean a worse outcome).
Time Frame: 4-month, 12-month, and 24-month time points (survey)
Population: The Early Childhood Oral Health 'Family' Impact scale score (range 0 - 16; higher scores mean a worse outcome)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oral Health Text Messages (OHT) | Child Wellness Text Messages (CWT)
Number analyzed (Participants) | 377 | 377
score on a scale
  24-month: number analyzed (Participants) | 272 | 270
  24-month | 1.03 (2.00) | 0.99 (1.80)
  12-month: number analyzed (Participants) | 282 | 290
  12-month | 1.14 (2.03) | 0.96 (1.79)
  4-month: number analyzed (Participants) | 290 | 288
  4-month | 0.65 (1.55) | 0.80 (1.76)

17. Secondary Outcome: Satisfaction With Text Message Program Features
Description: One item adapted from the Mobile App Rating Scale (MARS) to measure parent/caregiver participants' overall level of satisfaction with the text message program features (range 1 - 7; higher scores mean a better outcome).
Time Frame: 4-month time point (survey)
Population: Average level of satisfaction with text message program features (1='not satisfied at all', to 7='very much satisfied'; higher scores mean a better outcome)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oral Health Text Messages (OHT) | Child Wellness Text Messages (CWT)
Number analyzed (Participants) | 290 | 288
units on a scale | 6.12 (1.27) | 6.04 (1.35)

18. Secondary Outcome: Child Toothbrushing (Clinical Guidelines)
Description: An investigator-developed measure derived from the number of days and number of times parent/caregiver participants brushed or supervised brushing their child's teeth during a week recoded into "child met clinical guidelines for brushing" (brushing at least two times per day, seven days of the week) vs not.
Time Frame: 4-month, 12-month, and 24-month time points (survey)
Population: Number of parent/caregiver participants who indicated that they brushed or supervised brushing their child's teeth at least two times per day, seven days of the week.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Health Text Messages (OHT) | Child Wellness Text Messages (CWT)
Number analyzed (Participants) | 377 | 377
Participants
  24-Month: number analyzed (Participants) | 272 | 270
  24-Month | 177 | 147
  12-Month: number analyzed (Participants) | 282 | 290
  12-Month | 167 | 160
  4-Month: number analyzed (Participants) | 290 | 288
  4-Month | 214 | 156

19. Secondary Outcome: Parents/Caregivers Toothbrushing (Clinical Guidelines)
Description: An investigator-developed measure derived from the number of days and number of times parent/caregiver participants brushed their teeth during a week recoded into "parent/caregiver participants met clinical guidelines for brushing" (brushed at least two times per day, seven days of the week) vs not.
Time Frame: 4-month, 12-month, and 24-month time points (survey)
Population: Number of parent/caregiver participants who indicated that they brushed their teeth at least two times per day, seven days of the week.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Health Text Messages (OHT) | Child Wellness Text Messages (CWT)
Number analyzed (Participants) | 377 | 377
Participants
  24-Month: number analyzed (Participants) | 272 | 270
  24-Month | 188 | 175
  12-Month: number analyzed (Participants) | 282 | 290
  12-Month | 195 | 183
  4-Month: number analyzed (Participants) | 290 | 288
  4-Month | 208 | 191

20. Secondary Outcome: Diffusion of Text Messages (Satisfaction)
Description: One item adapted from the Mobile App Rating Scale (MARS) asks parent/caregiver participants whether they showed (or forwarded) text messages to anyone else
Time Frame: 4-month time point (survey)
Population: The iSmile study consisted of "oral health" text messages for parent/caregiver participants in the OHT arm, and "child wellness" text messages for parent/caregiver participants in the CWT arm. Diffusion of text messages assessed the number of parents/caregivers who showed (or forwarded) text messages to others.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Health Text Messages (OHT) | Child Wellness Text Messages (CWT)
Number analyzed (Participants) | 290 | 288
Participants | 168 | 177

21. Secondary Outcome: Text Message Program Star Rating
Description: One item adapted from the Mobile App Rating Scale (MARS) asks participants to give a star rating of the text message program. The star rating score range 1 star to 5 stars; a higher number of stars mean a better outcome.
Time Frame: 4-month time point (survey)
Population: The iSmile study consisted of "oral health" text messages for parent/caregiver participants in the OHT arm, and "child wellness" text messages for parent/caregiver participants in the CWT arm. The text message program star rating assessed the number of parent/caregiver participants who rated the text message program between 1 star and 5 stars.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Health Text Messages (OHT) | Child Wellness Text Messages (CWT)
Number analyzed (Participants) | 290 | 288
Participants
  1 star | 1 | 3
  2 stars | 12 | 7
  3 stars | 43 | 50
  4 stars | 89 | 88
  5 stars | 145 | 139
  prefer not to answer | 0 | 1

22. Secondary Outcome: Text Message Program Quality
Description: Parent/caregiver participants responded to an investigator developed survey to measure several aspects of text messages quality (range 1 - 7; higher scores mean a better outcome).
Time Frame: 4-month time point (survey)
Population: Parent/caregiver participants were asked 6 questions assessing the quality of the text messages (TMs) received during the program. Ratings were given on a 1 to 7 scale (higher scores mean a better outcome).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oral Health Text Messages (OHT) | Child Wellness Text Messages (CWT)
Number analyzed (Participants) | 290 | 288
units on a scale
  Relevant to cultural background | 5.81 (1.65) | 5.56 (1.71)
  Age appropriate for child | 6.0 (1.4) | 6.0 (1.4)
  Content of TMs easy to understand | 6.5 (1.1) | 6.6 (1.0)
  Easy to integrate into day/routine | 6.2 (1.2) | 6.2 (1.3)
  Language appropriate | 6.5 (1.1) | 6.5 (1.1)
  Relevant for you and your child | 6.2 (1.4) | 6.2 (1.4)

23. Other Pre Specified Outcome: Type of Beverage Consumed Between Meals
Description: Parent/caregiver participants are asked to indicate what beverage their child consumes most often between meals.
Time Frame: 4-month, 12-month, and 24-month time points (survey)
Population: Number of parent/caregiver participants indicating that their child consumed the beverage between meals.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Health Text Messages (OHT) | Child Wellness Text Messages (CWT)
Number analyzed (Participants) | 377 | 377
Participants
  24-Month: number analyzed (Participants) | 272 | 270
  24-Month: 1. Cow's milk | 31 | 31
  24-Month: 2. Juice or juice drinks | 63 | 77
  24-Month: 3. Diet soda pop or other sugar free beverages | 1 | 0
  24-Month: 4. Water | 164 | 149
  24-Month: 5. Regular soda pop or other sugared beverages | 1 | 1
  24-Month: 6. Flavored milk | 4 | 4
  24-Month: 7. Other | 3 | 2
  24-Month: Do not know | 2 | 1
  24-Month: Prefer not to answer | 3 | 5
  12-Month: number analyzed (Participants) | 282 | 290
  12-Month: 1. Cow's milk | 50 | 42
  12-Month: 2. Juice or juice drinks | 63 | 70
  12-Month: 3. Diet soda pop or other sugar free beverages | 1 | 0
  12-Month: 4. Water | 154 | 166
  12-Month: 5. Regular soda pop or other sugared beverages | 2 | 1
  12-Month: 6. Flavored milk | 4 | 4
  12-Month: 7. Other | 5 | 1
  12-Month: Do not know | 0 | 1
  12-Month: Prefer not to answer | 3 | 5
  4-Month: number analyzed (Participants) | 290 | 288
  4-Month: 1. Cow's milk | 48 | 56
  4-Month: 2. Juice or juice drinks | 63 | 69
  4-Month: 3. Diet soda pop or other sugar free beverages | 1 | 4
  4-Month: 4. Water | 159 | 147
  4-Month: 5. Regular soda pop or other sugared beverages | 3 | 0
  4-Month: 6. Flavored milk | 4 | 3
  4-Month: 7. Other | 6 | 7
  4-Month: Do not know | 2 | 1
  4-Month: Prefer not to answer | 4 | 1

24. Other Pre Specified Outcome: Challenge Week During the OHT Text Message Program
Description: We assessed the number of parent/caregiver participants in the OHT arm who agreed to do the challenge (setting the goal of brushing their child's teeth every day, twice per day) that occurred within the 4-month text message program.
Time Frame: 4-month time point
Population: Number of parent/caregiver participants in the OHT arm who agreed to do the challenge.
Measure: Count of Participants; unit: Participants
Arm/Group | OHT Group
Number analyzed (Participants) | 377
Participants
  Challenge one | 189
  Challenge two | 157

25. Other Pre Specified Outcome: Dental Caries (Per Subject)
Description: Number of primary teeth with new dental caries per child
Time Frame: 24-Month (oral health assessment)
Population: Number of primary teeth with new dental caries per child
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Health Text Messages (OHT) | Child Wellness Text Messages (CWT)
Number analyzed (Participants) | 160 | 156
Participants
  0 teeth with new caries | 91 | 95
  1 tooth with new caries | 19 | 15
  2 teeth with new caries | 13 | 16
  3 to 5 teeth with new caries | 22 | 16
  6 or more teeth with new caries | 15 | 14

ADVERSE EVENTS:
Time Frame: Up to 24 months
Arm/Group | Oral Health Text Messages (OHT) | Child Wellness Text Messages (CWT)
All-Cause Mortality (participants affected / at risk) | 1/377 | 0/377
Serious Adverse Events (participants affected / at risk) | 1/377 | 0/377
Other Adverse Events (participants affected / at risk) | 0/377 | 0/377
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Health Text Messages (OHT) (N=377) | Child Wellness Text Messages (CWT) (N=377)
Death - Probably not related to a study device (Social circumstances) | 1 | NA — Study team made a retention call for a follow-up survey on 10/14/20. A family member picked up and informed us that the parent/caregiver participant had died. No other details were disclosed. Study team ascertained that the death occurred 02/15/20.

LIMITATIONS AND CAVEATS:
Due to the COVID-19 pandemic, on March 12, 2020 Boston University Medical campus and Boston Medical Center IRB declared an immediate halt of in-person research activities. This resulted in a less than expected number of children attending the 12 and/or the 24 month oral health assessments.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-03-29): https://cdn.clinicaltrials.gov/large-docs/90/NCT03294590/Prot_SAP_001.pdf
  • Informed Consent Form (2019-03-29): https://cdn.clinicaltrials.gov/large-docs/90/NCT03294590/ICF_000.pdf